CLINICAL TRIAL: NCT03438266
Title: A Multicenter, Single-blind, Randomized, Controlled Study of the Safety and Effectiveness of JUVÉDERM VOLUMA® XC Injectable Gel for Cheek Augmentation Using Cannula
Brief Title: A Study of the Safety and Effectiveness of JUVÉDERM VOLUMA® XC Injectable Gel for Cheek Augmentation Using Cannula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1650-801-008
Record Dates: First submitted 2018-02-05; First posted 2018-02-19 (Actual); Results first posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Age-related Volume Deficit in the Mid-face
MeSH Terms: interventions — Cannula; Needles

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- JUVÉDERM VOLUMA® XC Injectable Gel with Cannula (Experimental): Participants had 1 cheek treated with JUVÉDERM VOLUMA® XC injectable gel with cannula.
  Interventions: Device: JUVÉDERM VOLUMA® XC injectable gel with cannula
- JUVÉDERM VOLUMA® XC Injectable Gel with Needle (Other): Participants had 1 cheek treated with JUVÉDERM VOLUMA® XC injectable gel with a needle.
  Interventions: Device: JUVÉDERM VOLUMA® XC injectable gel with needle

INTERVENTIONS:
Device: JUVÉDERM VOLUMA® XC injectable gel with cannula — Participants had 1 cheek treated with JUVÉDERM VOLUMA® XC injectable gel with cannula.
  Arms: JUVÉDERM VOLUMA® XC Injectable Gel with Cannula
Device: JUVÉDERM VOLUMA® XC injectable gel with needle — Participants had 1 cheek treated with JUVÉDERM VOLUMA® XC injectable gel with a needle.
  Arms: JUVÉDERM VOLUMA® XC Injectable Gel with Needle

SUMMARY:
The objective of this study is to evaluate the safety and effectiveness of JUVÉDERM VOLUMA® XC injectable gel using cannula in participants seeking correction of age-related volume deficit in the mid-face.

ELIGIBILITY:
Inclusion Criteria:

Male or female aged 35 to 65 (inclusive) years of age with overall mid-face severity of Moderate, Significant, or Severe for both cheeks on the Mid-Face Volume Deficit Scale (MFVDS);

Exclusion criteria:

* Has any facial procedures or trauma that may interfere with the study procedures and results;
* Has a history of anaphylaxis or allergy to lidocaine (or any amide-based anesthetics), hyaluronic acid (HA) products, or Streptococcal protein, or is planning to undergo allergen desensitization therapy during the term of the study;
* Has active autoimmune disease;
* Has current cutaneous or mucosal inflammatory or infectious processes.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-05-29 (Actual); Study Completion 2018-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Abrams, Study Director — Allergan
Locations (7):
- United States (7):
  - Skin Care and Laser Physicians of Beverly Hills, Los Angeles, California
  - Art of Skin MD, Solana Beach, California
  - Baumann Cosmetic and Research Institute, Miami, Florida
  - Saint Louis University Dermatology, St Louis, Missouri
  - Skin Laser & Surgery Specialists of NY/NJ, Hackensack, New Jersey
  - Rhoda S. Narins, MD, PC, White Plains, New York
  - Aesthetic Solutions, PA, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Additional information on study locations near you may be found at AllerganClinicalTrials.com. For any study not on AllerganClinicalTrials.com, please contact IR-CTRegistration@Allergan.com for assistance. — http://www.allerganclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 66 participants were enrolled in the study and 6 were excluded as screen failures. Only 60 participants were randomized and received study treatment.
Groups:
- JUVÉDERM VOLUMA® XC (All Participants): Participants had 1 cheek treated with JUVÉDERM VOLUMA® XC injectable gel with cannula and 1 cheek treated with JUVÉDERM VOLUMA® XC injectable gel with a needle.
Period: Overall Study
Arm/Group | JUVÉDERM VOLUMA® XC (All Participants)
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT) population included all randomized participants who received treatment with cannula on 1 cheek and treatment with needle on the contralateral (other) cheek.
Units Other Than Participants: Cheeks
Arm/Group | JUVÉDERM VOLUMA® XC (All Participants)
Number analyzed (Participants) | 60
Number analyzed (Cheeks) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.9 (6.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 59
  Black or African American | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 53

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mid-Face Volume Deficit Scale (MFVDS) Score
Description: The evaluating investigator (EI) assessed the participant's overall mid-face volume deficit for each cheek using a 6-point photonumeric scale, where: 0=None (moon face; fullness) [best] to 5=Severe (wasting) [worst]. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Screening) to Month 1
Population: mITT population included all randomized participants who received treatment with cannula on 1 cheek and treatment with needle on the contralateral (other) cheek.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JUVÉDERM VOLUMA® XC Injectable Gel With Cannula | JUVÉDERM VOLUMA® XC Injectable Gel With Needle
Number analyzed (Participants) | 60 | 60
score on a scale
  Baseline | 3.5 (0.62) | 3.5 (0.62)
  Change from Baseline at Month 1 | -1.8 (1.03) | -1.9 (0.96)
Statistical Analysis 1: Comparison: JUVÉDERM VOLUMA® XC Injectable Gel With Cannula vs JUVÉDERM VOLUMA® XC Injectable Gel With Needle; Change from Baseline at Month 1; Test type: Non-Inferiority — If the upper limit of the confidence interval at Month 1 was less than 0.5, then treatment with cannula was considered non-inferior to treatment with needle; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.05 to 0.25] — The 95% CI is based on the paired t-test

2. Secondary Outcome: Percentage of Participants With at Least a 1-Point Improvement (Decrease From Baseline) in MFVDS Score
Description: The EI assessed the participant's overall mid-face volume deficit for each cheek using a 6-point photonumeric scale, where: 0=None (moon face; fullness) [best] to 5=Severe (wasting) [worst]. The percentage of participants who showed ≥1-point improvement (decrease in severity) from Baseline is reported.
Time Frame: Baseline (Screening) to Month 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | JUVÉDERM VOLUMA® XC Injectable Gel With Cannula | JUVÉDERM VOLUMA® XC Injectable Gel With Needle
Number analyzed (Participants) | 60 | 60
percentage of participants | 93.3 [83.80 to 98.15] | 95.0 [86.08 to 98.96]
Statistical Analysis 1: Comparison: JUVÉDERM VOLUMA® XC Injectable Gel With Cannula vs JUVÉDERM VOLUMA® XC Injectable Gel With Needle; Test type: Other; Percentage Difference = -1.7, 95% CI 2-sided [-7.31 to 3.98]

3. Secondary Outcome: Change From Baseline in FACE-Q Satisfaction With Cheeks Questionnaire Score
Description: The participant completed the 5-item Satisfaction with Cheeks module of the FACE-Q questionnaire that evaluated various aspects of the cheeks including symmetry, smoothness, attractiveness, contour, and fullness using a 4-point scale where: 1=very dissatisfied to 4=very satisfied. The total score was transformed to a 0 to 100 point scale, with higher scores indicating greater satisfaction. A positive change from Baseline indicates improvement. The FACE-Q Satisfaction with Cheeks outcome was assessed by the participant overall and not by each cheek.
Time Frame: Baseline (Screening) to Month 1
Population: mITT population included all randomized participants who received treatment with cannula on 1 cheek and treatment with needle on the contralateral (other) cheek. FACE-Q is a global assessment and was administered per participant.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | JUVÉDERM VOLUMA® XC (All Participants)
Number analyzed (Participants) | 60
score on a scale
  Baseline | 32.1 (15.62)
  Change from Baseline at Month 1 | 55.5 (25.06)

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A TEAE is defined as an AE that initially occurred or increased in severity on or after the treatment start date.
Time Frame: Up to 3 months
Population: Safety population included all randomized participants who received at least 1 study treatment. The data for adverse events is reported by participant because both treatments were received at the same time and it included both treatment-related and non-treatment-related adverse events.
Measure: Count of Participants; unit: Participants
Arm/Group | JUVÉDERM VOLUMA® XC (All Participants)
Number analyzed (Participants) | 60
Participants | 7

ADVERSE EVENTS:
Time Frame: Up to 3 months
Description: The data for adverse events is reported by participant because both treatments were received at the same time and it included both treatment-related and non-treatment-related adverse events.
Arm/Group | JUVÉDERM VOLUMA® XC (All Participants)
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 3/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JUVÉDERM VOLUMA® XC (All Participants) (N=60)
Headache (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-10-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT03438266/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-13): https://cdn.clinicaltrials.gov/large-docs/66/NCT03438266/SAP_001.pdf